CLINICAL TRIAL: NCT02737280
Title: High Flow Humified Nasal Cannula Oxygen Therapy in Infants Younger Than 6 Months of Age With Viral Bronchiolitis Compared to Usual Oxygen Therapy : a Randomized Controlled Trial
Brief Title: High Flow Nasal Cannula Use in Infants With Bronchiolitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Marjo Renko, MD, PhD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EETTMK2015
Record Dates: First submitted 2016-02-26; First posted 2016-04-13 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Bronchiolitis
Keywords: infant; high flow nasal cannulae; oxygen therapy; bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual oxygen therapy (Active Comparator): Oxygen therapy with normal nasal cannula (for example MedKit Finland) 0-2 l/min
  Interventions: Device: MedKit Finland - Usual oxygen therapy
- High flow oxygen therapy (Experimental): High flow nasal cannula oxygen therapy with Airvo (TM, Fisher & Paykel Healthcare) device
  Interventions: Device: Airvo (TM, Fisher & Paykel Healthcare) - High flow oxygen therapy

INTERVENTIONS:
Device: Airvo (TM, Fisher & Paykel Healthcare) - High flow oxygen therapy — High flow nasal cannula therapy with Airvo (TM, Fisher & Paykel Healthcare) device
  Arms: High flow oxygen therapy
Device: MedKit Finland - Usual oxygen therapy — Oxygen therapy with normal nasal cannula (for example MedKit Finland) 0-2 l/min
  Arms: Usual oxygen therapy

SUMMARY:
Infants with viral bronchiolitis are currently treated with oxygen therapy if oxygen saturation is low. In earlier observational clinical studies, the use of high flow nasal cannulae therapy in infants with bronchiolitis has been associated with a decreased rate of intubation and intensive care. This study is a randomized controlled trial in two pediatric university hospitals in Finland comparing high flow nasal cannulae therapy to usual oxygen therapy in infants with bronchiolitis.

DETAILED DESCRIPTION:
Infants with viral bronchiolitis are currently treated with oxygen therapy if oxygen saturation is low. In earlier observational clinical studies, the use of high flow nasal cannulae therapy in infants with bronchiolitis has been associated with a decreased rate of intubation and intensive care. This study is a randomized controlled trial in five pediatric university hospitals in Finland comparing high flow nasal cannulae therapy to usual oxygen therapy in infants with bronchiolitis.

The investigators will recruit 160 infants who require oxygen therapy (oxygen saturation <92%) during hospitalization due to a viral bronchiolitis. The participants are randomized to receive oxygen therapy either with high flow or ordinary nasal cannula.The infants are closely observed by study physicians for clinical parameters. The primary end point is treatment failure (need for change of respiratory support method). Secondary endpoints are respiratory rate (RR) and oxygen saturation (%) at specific measuring points, time from randomisation to end of oxygen therapy and time from randomisation to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Admission to pediatric ward due to a presumed viral bronchiolitis
* Need of oxygen therapy (oxygen saturation < 92%)

Exclusion Criteria:

* Pertussis
* Needs intubation or CPAP on admission
* Severe congenital heart defect
* Down's syndrome

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment failure | 720 hours
  Treatment failure = need for change of respiratory support method

SECONDARY OUTCOMES:
Respiratory rate measured by the study physician/nurse | At 30 min, 60 min, 90 min, 4 hours, 8 hours
Oxygen saturation (%) | At 30 min, 60 min, 90 min, 4 hours, 8 hours
Time from randomisation to end of oxygen therapy | At 30 min, 60 min, 90 min, 4 hours, 8 hours
Time from hospital admission to discharge (hours) | 720 hours
  The date and time for admission and discharge will be registered for each participant and time from hospital admission to discharge is then calculated in hours and compared between the study groups.
Number of participants needing admission to intensive care unit (ICU) | 720 hours
  The number of participants needing admission to intensive care unit (ICU) will be registered in both treatment groups and that number divided by the total number of participants in the groups (percentages) are then compared between the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Marjo Renko, MD, PhD, Principal Investigator — University of Oulu
Locations (4):
- Finland (4):
  - Central Hospital Jyväskylä, Jyväskylä
  - Oulu Unversity Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: Undecided